CLINICAL TRIAL: NCT05483985
Title: Evaluation of the Alife Hera System as an Adjunctive Tool for the Prioritization of Embryos Deemed Suitable for Transfer: A Randomized Controlled Study
Brief Title: Evaluation of the Alife Hera System as an Adjunctive Tool for the Prioritization of Embryos Deemed Suitable for Transfer
Acronym: LOTUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alife Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP-01
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, 1:1 allocation in treatment and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Traditional Morphology (No Intervention): The embryo selection will be based on standard of care traditional morphology only.
- Device: Hera System (Experimental): For the Hera, the embryologist will use the consider both the standard morphology grade and the Hera System score on embryos that were already deemed suitable for transfer or freeze based on the standard morphology assessment to determine the most suitable embryo for transfer.
  Interventions: Device: Hera Score

INTERVENTIONS:
Device: Hera Score — The device uses patient metadata (patient age, day of image capture) and a software algorithm to analyze features of the blastocyst morphology to provide adjunctive information that may predict further development of the embryo to clinical pregnancy after embryo transfer.
  Arms: Device: Hera System

SUMMARY:
To evaluate the clinical pregnancy rate (pregnancy defined as fetal heartbeat at 6-8 weeks) with the adjunctive use of the Hera System (Hera System used with traditional morphological grading) with embryos already deemed suitable for transfer compared to trained embryologists using standard morphology criteria alone.

DETAILED DESCRIPTION:
To evaluate the clinical pregnancy rate (pregnancy defined as fetal heartbeat at 6-8 weeks) with the adjunctive use of the Hera System (Hera System used with traditional morphological grading) with embryos already deemed suitable for transfer compared to trained embryologists using standard morphology criteria alone.

To evaluate the performance and utilization of the Hera System as an adjunctive embryo grading and prioritization tool in an embryology lab setting with trained embryologists.

ELIGIBILITY:
Inclusion Criteria:

1. >21 and < 43 years of age
2. Women undergoing in vitro fertilization treatment using their own eggs
3. At least 8 eggs retrieved
4. Fertilization using only ejaculated sperm including donor sperm (fresh or frozen)
5. Single embryo transfer (SET)
6. Willing to comply with study protocol and procedures and be able to speak English
7. Willing to provide written informed consent

Exclusion Criteria:

1. Gestational carriers
2. Use of re-inseminated eggs
3. Use of donor eggs
4. History of cancer
5. Fertilization using surgically removed sperm
6. Transfer of multiple (more than one) embryos at once
7. Participants undergoing IVF with intent to bank embryos (i.e. no intention of embryo transfer for at least 6 months following egg retrieval)
8. Concurrent participation in another clinical study that might interfere with the study results in either study

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All women undergoing IVF
Enrollment: 440 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | up to 8 weeks
  The primary study endpoint is clinical pregnancy - defined as a fetal heartbeat at 6-8 weeks.

SECONDARY OUTCOMES:
Incidence of disagreement | week 1
  Incidence of disagreement for the top-ranked embryo between the Hera System and the embryologist.
User Experience | through study completion at 8 weeks
  Assessment of Hera System usability as reported by the embryologist using a user questionnaire.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - CCRM, Menlo Park, California
  - Reproductive Science Center, San Ramon, California
  - IVF Florida Reproductive Associates, Margate, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Ovation Fertility, Austin, Texas
  - Aspire Fertility, San Antonio, Texas
  - Reproductive Care Center, Sandy City, Utah